CLINICAL TRIAL: NCT04034056
Title: A Non-Interventional, Retrospective And Prospective, Multicenter, Single Arm Study Evaluating The Effectiveness And Safety Of Obinutuzumab In Patients With Previously Untreated Advanced Follicular Lymphoma
Brief Title: Untreated FolliculaR Lymphoma Treated With OBinituzumAb in a Non-interventional Study (URBAN)
Acronym: URBAN
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML41215
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — obinutuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Obinutuzumab
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — Induction phase: 1000 milligram (mg) intravenously (IV) on Day 1, 8, 15 of Cycle 1 an Day 1 of Cycles 2-6 or 2-8. Maintenance phase: 1000 mg IV every 2 months for 2 years or until disease progression (whatever occurs earlier).

SUMMARY:
To evaluate the effectiveness and safety of obinutuzumab in clinical routine in 1L FL measured by the % of relapse within 24 months from start of therapy.

DETAILED DESCRIPTION:
This observational study has been planned to evaluate the effectiveness of obinutuzumab in combination with chemotherapy in previously untreated advanced FL patients, in the real world setting in Italy. The study will allow to collect real-life data in a significant number of Italian patients when compared to participants in pivotal studies of obinutuzumab and thus will allow to verify in routine practice (after physician hands-on) the effectiveness and safety management in 50 reference sites all over the country.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent according to local regulations, after performing at least 2 cycles of induction treatment with Obinutuzumab and chemotherapy, within 1 year from beginning of treatment

Exclusion Criteria:

* Any contraindications to Obinutuzumab therapy according to local label for specific indication;
* Concomitant participation in an interventional clinical study;
* Participants not receiving treatment for untreated follicular lymphoma with Obinutuzumab according to standard of care and in line with local labeling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population taking part in the study will comprise patients aged ≥ 18 years in first treatment for advanced FL, in which Obinutuzumab are administered in combination with chemotherapy during the induction phase, followed by Obinutuzumab maintenance therapy. This indication and treatment scheme is that approved by the EMA as per EU countries agency and AIFA as per Italian local agency.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (46):
- Italy (46):
  - Ospedale Civile Dello Spirito Santo, Pescara, Abruzzo
  - AOU Policlinico Consorziale, Bari, Apulia
  - Giovanni Paolo II/I.R.C.C.S. Istituto Tumori, Bari, Apulia
  - Asl Bat Ospedale Mons. Dimiccoli, Barletta, Apulia
  - Ospedale Vito Fazzi, Lecce, Apulia
  - Casa Sollievo della Sofferenza U.O. Ematologia, San Giovanni Rotondo (FG), Apulia
  - Az. Osp. C. Panico, Tricase - LE, Apulia
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli, Reggio Calabria, Calabria
  - Azienda Ospedaliera S.G. Moscati, Avellino, Campania
  - A.O. S. Anna e San Sebastiano, Caserta, Campania
  - Istituto Nazionale Tumori Irccs Fondazione g. Pascale, Napoli, Campania
  - Ospedale Cardarelli, Napoli, Campania
  - Ospedale "A.Tortora" ? Ematologia, Pagani (Sa), Campania
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpigh, Bologna, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena, Modena, Emilia-Romagna
  - Az. Osp. Arcispedale S. Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO), Aviano, Friuli Venezia Giulia
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia, Udine, Friuli Venezia Giulia
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Lazio
  - Univesità La Sapienza Policlinico Umberto I, Rome, Lazio
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea-Universitr di Roma La Sapien, Rome, Lazio
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo, Lombardy
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - UOC Oncoematologia, Ospedale Maggiore Policlinico, Milano Policlinico Maggiore, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - Ospedale Di Circolo E Fondazione Macchi, Varese, Lombardy
  - Azienda Ospedaliera SS. Antonio E. Biagio E. Cesare Arrigo di Alessandria, Alessandria, Piedmont
  - Città della Salute e della Scienza di Torino. Presidio Molinette, Turin, Piedmont
  - Ospedale Businco, Cagliari, Sardinia
  - Osp. San Francesco, Nuoro, Sardinia
  - ARNAS Garibaldi, Catania, Sicily
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele, Catania, Sicily
  - Azienda Ospedaliera Vincenzo Cervello, Palermo, Sicily
  - Casa Di Cura La Maddalena, Palermo, Sicily
  - Ospedali Riuniti Umberto I, Ancona, The Marches
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - USL 4 di Prato - Nuovo Ospeale di Prato, Prato, Tuscany
  - A.O. Universitaria Senese, Siena, Tuscany
  - Azienda Ospedaliera S. Maria della Misericordia, Perugia, Umbria
  - Az. Osp. S. Maria, Terni, Umbria
  - Ematologia/immunologia Clinica Azienda Ospedaliera Policlinico di Padova, Padua, Veneto
  - Ospedale Ca Foncello, Treviso, Veneto
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Roma, Verona, Veneto

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Pinto A, Caltagirone M, Battista M, Gazzoli GC, Patti C, Pennese E, De Lorenzo S, Pavone V, Merli M, Chiarenza A, Gorgone AG, Piazza F, Puccini B, Noto A, Arcaini L, De Filippi R, Zinzani PL, Ferreri AJM, Ladetto M, Ferrari S, Gritti G. Exposure to obinutuzumab does not affect outcomes of SARS-CoV-2 infection in vaccinated patients with newly diagnosed advanced-stage follicular lymphoma. Br J Haematol. 2024 Dec;205(6):2219-2227. doi: 10.1111/bjh.19661. Epub 2024 Jul 22. PMID 39039666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 299 participants with untreated advanced follicular lymphoma (FL) took part in the study at 50 investigative sites in Italy from 02 September 2019 to 22 April 2024.
Pre-assignment Details: This was a prospective and retrospective data collection study. Participants were observed for safety and efficacy of obinutuzumab during the 6-month induction treatment with obinutuzumab and chemotherapy, and 24-month maintenance treatment with obinutuzumab monotherapy followed by 1 year of follow up.
Groups:
- Obinutuzumab: Participants who received at least 2 cycles of obinutuzumab and chemotherapy as IV infusion as induction treatment, followed by obinutuzumab monotherapy as maintenance treatment per physician's decision in accordance with local clinical practice and local labelling were observed for efficacy and safety for up to 3.5 years or until PD, withdrawal of consent, study termination by sponsor or death, whichever occurred first (1 cycle = 28 days).
Period: Overall Study
Arm/Group | Obinutuzumab
Started | 299
Completed | 228
Not Completed | 71
Not completed — Withdrawal by Subject | 2
Not completed — Reason Not Specified | 13
Not completed — Adverse Event | 56

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were enrolled in the study.
  Data for Race and Ethnicity was not collected.
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158
  Male | 141
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression of Disease at Year 2 (POD24)
Description: POD24=time from date of treatment initiation with obinutuzumab until first documented PD/death due to PD, whichever occurs first, within 24 months from start of treatment with obinutuzumab. According to standard Cheson criteria & Deauville 5-point scale, PD=20% increase in sum of longest diameters (LD) of target lesions; for small lymph nodes measuring <15 millimeters (mm) post therapy, a minimum absolute increase of 5 mm & LD should exceed 15 mm; appearance of a new lesion; any bone marrow involvement & any 18F-fluorodeoxyglucose-positron emission tomography (FDG-PET) results. Participants with no PD & who didn't die due to PD/were lost to follow-up at time of analysis were censored at date of last tumor assessment where no progression was documented/last date of follow-up for disease, whichever was last. Participants without post-baseline tumor assessments were censored at time of their baseline visit unless death due to PD occurred prior to their first scheduled tumor assessment.
Time Frame: At Year 2
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab. Overall number analyzed is the number of participants with data available for POD24 analysis. Percentages have been rounded off.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 281
percentage of participants | 8.9 [5.8 to 12.9]

2. Secondary Outcome: Percentage of Participants With Progression-free Survival at Year 2 (PFS2)
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. According to standard Cheson criteria and Deauville 5-point scale, PD was defined as 20% increase in the sum of LD of target lesions; for small lymph nodes measuring < 15 mm post-therapy, a minimum absolute increase of 5 mm and the LD should exceed 15 mm; the appearance of a new lesion; any bone marrow involvement and any FDG-PET results. Kaplan-Meier estimate of the PFS2 rate at 2 years (that is, the estimated percentage of participants with PFS2 at Year 2) is presented.
Time Frame: At Year 2
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab. Percentages have been rounded off.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Obinutuzumab: Participants who received at least 2 cycles of obinutuzumab and chemotherapy as IV infusion as induction treatment, followed by obinutuzumab monotherapy as maintenance treatment per physician's decision in accordance with local clinical practice and local labelling were observed for efficacy and safety for up to 3.5 years or until PD, withdrawal of consent, study termination by sponsor or death, whichever occured first (1 cycle = 28 days).
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
percentage of participants | 85.6 [81.1 to 89.4]

3. Secondary Outcome: Percentage of Participants With PFS at Year 3 (PFS3)
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. According to standard Cheson criteria and Deauville 5-point scale, PD was defined as 20% increase in the sum of LD of target lesions; for small lymph nodes measuring < 15 mm post therapy, a minimum absolute increase of 5 mm and the LD should exceed 15 mm; appearance of a new lesion; any bone marrow involvement & any FDG-PET results. Kaplan-Meier estimate of the PFS3 rate at 3 years (that is, the estimated percentage of participants with PFS3 at Year 3) is presented.
Time Frame: At Year 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
percentage of participants | 76.6 [71.4 to 81.3]

4. Secondary Outcome: Time to Next Treatment (TTNT)
Description: TTNT was defined as the time to initiation of subsequent systemic anti-cancer therapy following initiation of obinutuzumab containing therapy. Participants who did not start subsequent systemic anti-cancer therapy were censored at the date of the last study visit.
Time Frame: Up to approximately 56 months
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab.
Measure: Median (Full Range); unit: days
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
days | 1118 [167 to 1478]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from initiation of study treatment to death from any cause. Participants who were still alive at the time of analysis and participants who were lost to follow-up were censored at their last time known to be alive.
Time Frame: Up to approximately 56 months
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
days | 1269 [1135 to 1277]

6. Secondary Outcome: Time From First Dose to Loss of Clinical Benefit (TTLCB)
Description: TTLCB was defined as the time from first dose to loss of clinical benefit as assessed by the treating physician (single or multiple reasons possible: e.g. PD, deterioration in Eastern Cooperative Oncology Group Performance Status (ECOG PS), death, other). Participants who did not lose clinical benefit were censored at the date of the last study visit. Participants without post-baseline tumor assessments were censored at the time of their baseline visit unless death occurred prior to their first scheduled tumor assessment.
Time Frame: Up to approximately 56 months
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab.
Measure: Median (Full Range); unit: days
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
days | 1127 [167 to 1266]

7. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a complete response (CR) or partial response (PR) at mid and end of induction (6 months), and during and after maintenance therapy (24 months), as per clinical practice, with and without FDG-PET. Per standard Cheson criteria and Deauville 5-point scale, CR was defined as complete disappearance of all target lesions & all nodes with long axis < 10 mm or ≥ 30% decrease in sum of LD of target lesions with normalization of FDG-PET (Deauville score 1-3); no new lesions & no bone marrow involvement. PR was defined as ≥ 30% decrease in sum of LD of target lesions but not a CR; positive FDG-PET (Deauville score 4-5); no new lesions and any bone marrow involvement. The Deauville 5-Point Scale is based on visual interpretation of FDG uptake. Scale ranges from 1 to 5, where 1 (best)=no FDG uptake; 2=FDG uptake ≤ mediastinum; 3=FDG uptake > mediastinum but ≤ liver; 4=FDG uptake moderately > liver; 5 (worst)=FDG uptake markedly > than liver.
Time Frame: Up to approximately 56 months
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab. Number analyzed per timepoint are unique number of participants out of all the assessed participants with data available for analysis at the specified timepoint. Different participants may have contributed data for each timepoint. Percentages have been rounded off.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
percentage of participants
  During Induction: number analyzed (Participants) | 220
  During Induction | 95 [91.2 to 97.5]
  End of Induction: number analyzed (Participants) | 271
  End of Induction | 95.6 [92.4 to 97.7]
  During Maintenance: number analyzed (Participants) | 220
  During Maintenance | 93.6 [89.6 to 96.5]
  End of Maintenance: number analyzed (Participants) | 159
  End of Maintenance | 94.3 [89.5 to 97.4]

8. Secondary Outcome: Percentage of Participants With CR
Description: According to standard Cheson criteria and Deauville 5-point scale, CR was defined as complete disappearance of all target lesions and all nodes with long axis < 10 mm or ≥ 30% decrease in the sum of LD of target lesions with normalization of FDG-PET (Deauville score 1-3); no new lesions and no bone marrow involvement. CR was assessed at mid and end of induction (6 months), and during and after maintenance therapy (24 months), as per clinical practice, with and without FDG-PET results. The Deauville 5-Point Scale is based on visual interpretation of FDG uptake. Scale ranges from 1 to 5, where 1 (best)=no FDG uptake; 2=FDG uptake ≤ mediastinum; 3=FDG uptake > mediastinum but ≤ liver; 4=FDG uptake moderately > liver; 5 (worst)=FDG uptake markedly > than liver.
Time Frame: Up to approximately 56 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
percentage of participants
  During Induction: number analyzed (Participants) | 220
  During Induction | 35.9 [29.6 to 42.6]
  End of Induction: number analyzed (Participants) | 271
  End of Induction | 79.7 [74.4 to 84.3]
  During Maintenance: number analyzed (Participants) | 220
  During Maintenance | 87.7 [82.6 to 91.8]
  End of Maintenance: number analyzed (Participants) | 159
  End of Maintenance | 90.6 [84.9 to 94.6]

9. Secondary Outcome: Percentage of Participants With CR at 30 Months (CR30)
Description: According to standard Cheson criteria and Deauville 5-point scale, CR at 30 months was defined as complete disappearance of all target lesions and all nodes with long axis < 10 mm or ≥ 30% decrease in the sum of LD of target lesions with normalization of FDG-PET (Deauville score 1-3); no new lesions and no bone marrow involvement. The Deauville 5-Point Scale is based on visual interpretation of FDG uptake. Scale ranges from 1 to 5, where 1 (best)=no FDG uptake; 2=FDG uptake ≤ mediastinum; 3=FDG uptake > mediastinum but ≤ liver; 4=FDG uptake moderately > liver; 5 (worst)=FDG uptake markedly > than liver.
Time Frame: At 30 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
percentage of participants | 91 [87.1 to 94]

10. Secondary Outcome: Duration of Response (DOR)
Description: DOR=time from first documentation of CR/PR until PD, as evaluated by physician according to routine clinical practice/death. CR=complete disappearance of all target lesions & all nodes with long axis <10 mm/ ≥30% decrease in sum of LD of target lesions with normalization of FDG-PET (Deauville score 1-3); no new lesions & no bone marrow involvement. PR= ≥30% decrease in sum of LD of target lesions but not CR; positive FDG-PET (Deauville score 4-5); no new lesions & any bone marrow involvement. PD=20% increase in sum of LD of target lesions; for small lymph nodes measuring <15 mm post therapy, minimum absolute increase of 5 mm & LD should exceed 15 mm; appearance of new lesion; any bone marrow involvement & FDG-PET results. Deauville 5-Point Scale is based on visual interpretation of FDG uptake. Scale ranges from 1-5, where 1 (best)=no FDG uptake; 2=FDG uptake ≤mediastinum; 3=FDG uptake >mediastinum but ≤liver; 4=FDG uptake moderately >liver; 5 (worst)=FDG uptake markedly >than liver.
Time Frame: Up to approximately 56 months
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab. Overall number analyzed included participants with OR i.e responders. Different participants with responses at different timepoints during the study may have contributed to the summarized data.
Measure: Median (Full Range); unit: days
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 293
days | 1010 [73 to 1168]

11. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as time from first dose of obinutuzumab to first documented response (CR or PR) as assessed in clinical routine. Per standard Cheson criteria & Deauville 5-point scale, CR was defined as the complete disappearance of all target lesions and all nodes with long axis < 10 mm or ≥ 30% decrease in the sum of LD of target lesions with normalization of FDG-PET (Deauville score 1-3); no new lesions and no bone marrow involvement. PR was defined as ≥30% decrease in the sum of LD of target lesions but not a CR (Deauville score 4-5); no new lesions & any bone marrow involvement. The Deauville 5-Point Scale is based on visual interpretation of FDG uptake. Scale ranges from 1 to 5, where 1 (best)=no FDG uptake; 2=FDG uptake ≤ mediastinum; 3=FDG uptake > mediastinum but ≤ liver; 4=FDG uptake moderately > liver; 5 (worst)=FDG uptake markedly > than liver.
Time Frame: Up to approximately 56 months
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab.
Measure: Median (Full Range); unit: days
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
days | 96 [15 to 577]

12. Secondary Outcome: Percentage of Participants With SD
Description: According to standard Cheson criteria and Deauville 5-point scale, SD was defined as < 10% decrease or ≤ 20% increase in the sum of LD of target lesions; no new lesions; any bone marrow involvement and any FDG-PET results. SD was assessed at mid and end of induction (6 months), and during and after maintenance therapy (24 months).
Time Frame: Up to approximately 56 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
percentage of participants
  During Induction: number analyzed (Participants) | 220
  During Induction | 2.3 [0.7 to 5.2]
  End of Induction: number analyzed (Participants) | 271
  End of Induction | 1.5 [0.4 to 3.7]
  During Maintenance: number analyzed (Participants) | 220
  During Maintenance | 2.3 [0.7 to 5.2]
  End of Maintenance: number analyzed (Participants) | 159
  End of Maintenance | 1.9 [0.4 to 5.4]

13. Secondary Outcome: Percentage of Participants With FDG-PET Response at End of Induction and End of Maintenance
Description: ORR was defined as percentage of participants with a CR/PR at end of induction & maintenance therapy, as per clinical practice, with FDG-PET. According to standard Cheson criteria & Deauville 5-point scale, CR was defined as complete disappearance of all target lesions & all nodes with long axis < 10 mm or ≥ 30% decrease in sum of LD of target lesions with normalization of FDG-PET (Deauville score 1-3); no new lesions & no bone marrow involvement. PR was defined as ≥30% decrease in sum of LD of target lesions but not a CR; positive FDG-PET (Deauville score 4-5); no new lesions & any bone marrow involvement. The Deauville 5-Point Scale is based on visual interpretation of FDG uptake. Scale ranges from 1 to 5, where 1 (best)=no FDG uptake; 2=FDG uptake ≤ mediastinum; 3=FDG uptake > mediastinum but ≤ liver; 4=FDG uptake moderately > liver; 5 (worst)=FDG uptake markedly > than liver.
Time Frame: Up to approximately 56 months
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
percentage of participants
  End of Induction: number analyzed (Participants) | 271
  End of Induction | 95.6 [92.4 to 97.7]
  End of Maintenance: number analyzed (Participants) | 159
  End of Maintenance | 94.3 [89.5 to 97.4]

14. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 185 days after the final obinutuzumab dose or until initiation of another anti-cancer therapy (approximately 48 months)
Population: Safety population included all participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
Participants | 287

15. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any AE that meets any of the following criteria: is fatal; life-threatening; requires or prolongs inpatient hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study medicine and is a significant medical event in the physician's judgment.
Time Frame: as for outcome 14
Population: Safety population included all participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
Participants | 121

16. Secondary Outcome: Number of Participants With Adverse Events of Special Interests (AESIs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AESIs for this study may include the following: tumor lysis syndrome (TLS), irrespective of causality; second malignancies; cases of potential medicine-induced liver injury that include an elevated alanine aminotransferase (ALT) or aspartate transaminase (AST) in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's law and suspected transmission of an infectious agent by the study medicine.
Time Frame: as for outcome 14
Population: Safety population included all participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
Participants | 9

17. Secondary Outcome: Number of Participants With Infusion-related Reactions (IRRs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. IRRs were defined as all AEs that occurred during or within 24 hours after study treatment infusion and were judged to be related to infusion of study treatment.
Time Frame: as for outcome 14
Population: Safety population included all participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 299
Participants | 38

18. Secondary Outcome: Percentage of Participants With PFS2 Stratified by Follicular Lymphoma International Prognostic Index (FLIPI)
Description: PFS=time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. Per standard Cheson criteria & Deauville 5-point scale, PD=20% increase in sum of LD of target lesions; for small lymph nodes measuring <15 mm post-therapy, a minimum absolute increase of 5 mm & the LD should exceed 15 mm; appearance of a new lesion; any bone marrow involvement & any FDG-PET results. The FLIPI tool predicts the prognosis of participants diagnosed with FL. Prognosis depends on 5 FLIPI risk factors: age >60 years, Ann Arbor stage III-IV, hemoglobin (Hb) level <12 grams per deciliter (gm/dL), >4 nodal areas & raised lactate dehydrogenase (LDH) levels. Each factor was given a point if it was positive. FLIPI score range from 0-5 where 0-1 = low risk; 2=intermediate risk and 3-5=high risk. Higher score indicates worse prognosis. Participants who were event-free at 2 years, stratified by FLIPI score are presented.
Time Frame: At Year 2
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab. Overall number analyzed is the number of participants who were progression-free at 2 years and were evaluable for this outcome measure. Percentages have been rounded off.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 254
percentage of participants
  FLIPI Score 0 | 0
  FLIPI Score 1 | 6.3
  FLIPI Score 2 | 37.4
  FLIPI Score 3 | 40.6
  FLIPI Score 4 | 12.6
  FLIPI Score 5 | 3.1

19. Secondary Outcome: Percentage of Participants With PFS2 Stratified by ECOG PS
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. PD was defined as outlined in the description of outcome measure 1 (POD24). ECOG-PS assessed participant's performance status on a 5 point scale where 0=fully active, able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, but ambulatory, able to carry out light/sedentary work; 2=ambulatory, capable of all self-care, but unable to carry out any work activities (>50% of waking hours); 3=capable of only limited self-care, confined to bed/chair (>50% of waking hours); 4=completely disabled, cannot carry on any selfcare, totally confined to bed or chair and 5=Dead. Higher score=lower performance. Data for participants who were event-free at 2 years, stratified by ECOG-PS score are presented.
Time Frame: At Year 2
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 142
percentage of participants
  ECOG PS Score 0 | 55.6
  ECOG PS Score 1 | 40.8
  ECOG PS Score 2 | 2.8
  ECOG PS Score 3 | 0.7
  ECOG PS Score 4 | 0
  ECOG PS Score 5 | 0

20. Secondary Outcome: Percentage of Participants With PFS2 Stratified by Age
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. According to standard Cheson criteria and Deauville 5-point scale, PD was defined as 20% increase in the sum of LD of target lesions; for small lymph nodes measuring < 15 mm post-therapy, a minimum absolute increase of 5 mm and the LD should exceed 15 mm; the appearance of a new lesion; any bone marrow involvement and any FDG-PET results. Data for participants who were event-free at 2 years, stratified by age (≤60 years & >60 years) are presented.
Time Frame: At Year 2
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 256
percentage of participants
  ≤ 60 Years | 44.5
  > 60 Years | 55.5

21. Secondary Outcome: Percentage of Participants With PFS2 Stratified by Chemotherapy Backbone Choice
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. According to standard Cheson criteria and Deauville 5-point scale, PD was defined as 20% increase in the sum of LD of target lesions; for small lymph nodes measuring < 15 mm post-therapy, a minimum absolute increase of 5 mm and the LD should exceed 15 mm; the appearance of a new lesion; any bone marrow involvement and any FDG-PET results. Participants treated with chemotherapy were given the following options: Bendamustine; CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone), and CVP (cyclophosphamide, vincristine, prednisone). Data for participants who were event-free at 2 years, stratified by chemotherapy backbone are presented.
Time Frame: At Year 2
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 256
percentage of participants
  Bendamustine | 47.3
  CHOP | 47.3
  CVP | 5.5

22. Secondary Outcome: Percentage of Participants With PFS2 Stratified by Hepatitis B Virus (HBV) Infection
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. According to standard Cheson criteria and Deauville 5-point scale, PD was defined as 20% increase in the sum of LD of target lesions; for small lymph nodes measuring < 15 mm post-therapy, a minimum absolute increase of 5 mm and the LD should exceed 15 mm; the appearance of a new lesion; any bone marrow involvement and any FDG-PET results. History of past/resolved infection or latent HBV after prophylaxis as per standard treatment guidelines was assessed. Data for participants who were event-free at 2 years, stratified by positive & negative HBV infection are presented.
Time Frame: At Year 2
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 230
percentage of participants
  Positive HBV | 4.3
  Negative HBV | 95.7

23. Secondary Outcome: Percentage of Participants With PFS2 Stratified by Presence of Autoimmune Disease, Renal and Hepatobilliary Disorders
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. According to standard Cheson criteria and Deauville 5-point scale, PD was defined as 20% increase in the sum of LD of target lesions; for small lymph nodes measuring < 15 mm post-therapy, a minimum absolute increase of 5 mm and the LD should exceed 15 mm; the appearance of a new lesion; any bone marrow involvement and any FDG-PET results. Data for participants who were event-free at 2 years, stratified by a history of autoimmune, renal and hepatobilliary disorders are presented.
Time Frame: At Year 2
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 206
percentage of participants
  Immune System Disorders | 7
  Hepatobilliary Disorders | 9.8
  Renal Disorders | 4.3

24. Secondary Outcome: Percentage of Participants With PFS3 Stratified by FLIPI
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. Per standard Cheson criteria & Deauville 5-point scale, PD was defined as 20% increase in sum of LD of target lesions; for small lymph nodes measuring <15 mm post-therapy, a minimum absolute increase of 5 mm & the LD should exceed 15 mm; appearance of a new lesion; any bone marrow involvement & any FDG-PET results. The FLIPI tool predicts the prognosis of participants diagnosed with FL. Prognosis depends on 5 FLIPI risk factors: age >60 years, Ann Arbor stage III-IV, Hb level <12 gm/dL, >4 nodal areas & raised LDH levels. Each factor was given a point if it was positive. FLIPI score range from 0-5 where 0-1 = low risk; 2=intermediate risk and 3-5=high risk. Higher score indicates worse prognosis. Participants who were event-free at 3 years, stratified by FLIPI score are presented.
Time Frame: At Year 3
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab. Overall number analyzed is the number of participants who were progression-free at 3 years and were evaluable for this outcome measure. Percentages have been rounded off.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 227
percentage of participants
  FLIPI Score 0 | 0
  FLIPI Score 1 | 5.3
  FLIPI Score 2 | 39.6
  FLIPI Score 3 | 40.5
  FLIPI Score 4 | 11.5
  FLIPI Score 5 | 3.1

25. Secondary Outcome: Percentage of Participants With PFS3 Stratified by ECOG PS
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. PD was defined as outlined in the description of outcome measure 1 (POD24). ECOG-PS assessed participant's performance status on a 5 point scale where 0=fully active, able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, but ambulatory, able to carry out light/sedentary work; 2=ambulatory, capable of all self-care, but unable to carry out any work activities (>50% of waking hours); 3=capable of only limited self-care, confined to bed/chair (>50% of waking hours); 4=completely disabled, cannot carry on any selfcare, totally confined to bed or chair and 5=Dead. Higher score=lower performance. Data for participants who were event-free at 3 years, stratified by ECOG-PS score are presented.
Time Frame: At Year 3
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 126
percentage of participants
  ECOG PS Score 0 | 57.1
  ECOG PS Score 1 | 39.7
  ECOG PS Score 2 | 3.2
  ECOG PS Score 3 | 0
  ECOG PS Score 4 | 0
  ECOG PS Score 5 | 0

26. Secondary Outcome: Percentage of Participants With PFS3 Stratified by Age
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. According to standard Cheson criteria and Deauville 5-point scale, PD was defined as 20% increase in the sum of LD of target lesions; for small lymph nodes measuring < 15 mm post-therapy, a minimum absolute increase of 5 mm and the LD should exceed 15 mm; the appearance of a new lesion; any bone marrow involvement and any FDG-PET results. Data for participants who were event-free at 3 years, stratified by age (≤60 years & >60 years) are presented.
Time Frame: At Year 3
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 229
percentage of participants
  ≤ 60 Years | 46.3
  > 60 Years | 53.7

27. Secondary Outcome: Percentage of Participants With PFS3 Stratified by Chemotherapy Backbone Choice
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. According to standard Cheson criteria and Deauville 5-point scale, PD was defined as 20% increase in the sum of LD of target lesions; for small lymph nodes measuring < 15 mm post-therapy, a minimum absolute increase of 5 mm and the LD should exceed 15 mm; the appearance of a new lesion; any bone marrow involvement and any FDG-PET results. Participants treated with chemotherapy were given the following options: Bendamustine; CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone), and CVP (cyclophosphamide, vincristine, prednisone). Data for participants who were event-free at 3 years, stratified by chemotherapy backbone are presented.
Time Frame: At Year 3
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 229
percentage of participants
  Bendamustine | 45.4
  CHOP | 48.9
  CVP | 5.7

28. Secondary Outcome: Percentage of Participants With PFS3 Stratified by HBV Infection
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. According to standard Cheson criteria and Deauville 5-point scale, PD was defined as 20% increase in the sum of LD of target lesions; for small lymph nodes measuring < 15 mm post-therapy, a minimum absolute increase of 5 mm and the LD should exceed 15 mm; the appearance of a new lesion; any bone marrow involvement and any FDG-PET results. History of past/resolved infection or latent HBV after prophylaxis as per standard treatment guidelines was assessed. Data for participants who were event-free at 3 years, stratified by positive & negative HBV infection are presented.
Time Frame: At Year 3
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 205
percentage of participants
  Positive HBV | 4.4
  Negative HBV | 95.6

29. Secondary Outcome: Percentage of Participants With PFS3 Stratified by Presence of Autoimmune Disease, Renal and Hepatobilliary Disorders
Description: PFS was defined as the time from the date of treatment initiation until the first documented PD measured by routine clinical care or death from any cause, whichever occurred first. According to standard Cheson criteria and Deauville 5-point scale, PD was defined as 20% increase in the sum of LD of target lesions; for small lymph nodes measuring < 15 mm post-therapy, a minimum absolute increase of 5 mm and the LD should exceed 15 mm; the appearance of a new lesion; any bone marrow involvement and any FDG-PET results. Data for participants who were event-free at 3 years, stratified by a history of autoimmune, renal and hepatobilliary disorders are presented. Percentages have been rounded off.
Time Frame: At Year 3
Population: Efficacy population included all participants who were enrolled and received at least two cycles of obinutuzumab. Overall number analyzed is the number of participants who were progression-free at 3 years and were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 182
percentage of participants
  Immune System Disorders | 7.4
  Hepatobilliary Disorders | 8.7
  Renal Disorders | 4.4

ADVERSE EVENTS:
Time Frame: All cause mortality: Up to 56 months SAEs and non-serious AEs: Up to 185 days after the final obinutuzumab dose or until initiation of another anti-cancer therapy, whichever occurred first (approximately 48 months)
Description: Safety population included all participants who were enrolled in the study.
Arm/Group | Obinutuzumab
All-Cause Mortality (participants affected / at risk) | 54/299
Serious Adverse Events (participants affected / at risk) | 121/299
Other Adverse Events (participants affected / at risk) | 113/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab (N=299)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Lymphoma (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (5)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Dyspnoea (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pulmonary oedema (Cardiac disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Adenocarcinoma of colon (Gastrointestinal disorders) | 2 (2)
Colon cancer (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Cholangiocarcinoma (Hepatobiliary disorders) | 1 (1)
Interstitial lung disease (Immune system disorders) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 51 (55)
COVID-19 pneumonia (Infections and infestations) | 25 (31)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 11 (11)
Post-acute COVID-19 syndrome (Infections and infestations) | 1 (1)
Psoas abscess (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Acute respiratory failure (Metabolism and nutrition disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Monoplegia (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Renal stone removal (Surgical and medical procedures) | 1 (1)
Ureteric calculus removal (Surgical and medical procedures) | 1 (1)
Uterine polypectomy (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab (N=299)
Neutropenia (Blood and lymphatic system disorders) | 113 (221)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-05-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT04034056/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT04034056/SAP_001.pdf